CLINICAL TRIAL: NCT06375382
Title: Effects of Acupuncture on Abdominal Pain-related Intestinal Flora in Patients With Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYS2024-01
Record Dates: First submitted 2024-03-31; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Gastrointestinal Microbiome; Abdominal Pain; Acupuncture
MeSH Terms: conditions — Crohn Disease; Abdominal Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): Receiving acupuncture and moxibustion
  Interventions: Other: acupuncture
- sham acupuncture group (Sham Comparator): Receiving sham acupuncture and sham moxibustion
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: acupuncture — We selected acupoints including Zhongwan (CV12) and bilateral Shangjuxu (ST37), Sanyinjiao (SP6), Gongsun (SP4), Taichong (LR3), Taixi (KI3), Hegu (LI4), and Quchi (LI11)17 according to the World Health Organization standard. Single-use 0.30×40 mm or 0.30×25 mm acupuncture needles (Hwato, Suzhou, China) 27,28 were vertically inserted into each acupoint to 20-30 mm depth to obtain a deqi sensation (a soreness, distention, numbness or heaviness sensation). Bilateral Zusanli (ST36) and Tianshu (ST25) were selected for moxibustion. Pure moxa sticks (diameter: 2.8 cm; Hanyi, Nanyang, China) were ignited and fixed on a moxibustion stand at a distance of 3-5 cm to the surface of acupoints. The temperature of skin surface at the acupoints was maintained at 43 ± 1°C and monitored with a miniature infrared thermometer (Fluke 62, Fluke Corporation, Everett, WA, USA). Acupuncture and moxibustion were concomitantly performed for 30 min.
  Arms: acupuncture group
Other: Sham acupuncture — Sham acupuncture needles (0.35×40 mm) with flat tips (Hwato, Suzhou, China) were inserted towards the same acupoints to induce slight pain but without penetrating the skin. Sham moxibustion was made by igniting the same type of moxa sticks but fixing them at a distance of 8-10 cm from the skin of acupoints to maintain the temperature at 37 ± 1°C. Sham acupuncture and moxibustion were concomitantly performed for 30 min.
  Arms: sham acupuncture group

SUMMARY:
Crohn's disease is an intestinal inflammatory disease, causing abdominal pain, diarrhea and other symptoms. The intestinal flora disorder is closely related to the occurrence and development of Crohn's disease. Acupuncture can induce remission of Crohn's disease during mild to moderate active period, improve clinical symptoms such as abdominal pain. This study is to screen the intestinal bacteria related to abdominal pain in CD, and explore the effects of acupuncture on the intestinal flora related to abdominal pain in CD patients.

DETAILED DESCRIPTION:
1. to screen the intestinal flora associated with CD abdominal pain.
2. to explore the effects of acupuncture and on abdominal pain and abdominal pain related intestinal flora in CD patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75, no gender limit;
2. disease in mild and moderate active period: 150≤CDAI<450 and meet at least one of the following: serum C-reactive protein (CRP) levels ≥5mg/L, Fecal calprotectin concentration≥250μg/g or endoscopic examination shows ulcers. remission period: CDAI <150 and meet at least one of the following: serum CRP<5 mg/L, Fecal calprotectin concentration <250μg/g or endoscopic examination shows no ulcer;
3. patients were not taking medication or were only taking one or more of the following drugs: mesalazine (≤4g/d and mesalazine was used for at least 1 month), prednisone (≤15mg/d and prednisone was used for at least 1 month) and / or azathioprine (≤1mg/kg/d and azathioprine was used for at least 3 month);
4. those who have not used biologics within 3 months before entering the study;
5. those who have never experienced acupuncture;
6. those who understand and agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. patients who are recently pregnant or in pregnancy or lactation;
2. patients with serious organic diseases;
3. patients diagnosed as psychosis;
4. patients who suffer from multiple diseases and need to take other drugs for a long time, and may affect the observation of the efficacy of this trial;
5. severe skin diseases (such as erythema nodosum, pyoderma gangrenosum, etc.), eye diseases (such as iritis, uveitis, etc.), thromboembolic diseases and other serious extraintestinal manifestations;
6. there are serious intestinal fistula, abdominal abscess, intestinal stenosis and obstruction, perianal abscess, gastrointestinal hemorrhage, intestinal perforation and other complications;
7. patients with short bowel syndrome who have undergone abdominal or gastrointestinal surgery in the past half a year;
8. there are skin diseases or defects in the selected area of acupuncture and moxibustion that cannot be performed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Abdominal pain remission rate | Week 12
  The abdominal pain relief rate is the ratio of the number of subjects with abdominal pain relief at the end of 12 weeks of treatment to the total number of subjects.

SECONDARY OUTCOMES:
Crohn's disease activity index （CDAI） | Week 12
  Between-group assessment by difference in Crohn's Disease Activity Index (CDAI) at 12 weeks from baseline. The minimum value is 0 and there is no upper limit. 0-150: disease in remission; 151-220: mild active disease; 221-450: moderate active disease; values above 450: severe active disease. Higher scores mean a worse outcome.
Hospital anxiety and depression scale (HADS) | Week 12
  Difference in Hospital anxiety and depression scale (HADS) scores from baseline at 12 weeks was used for between-group assessment. The minimum score is 0, and the maximum score is 21. Higher scores mean a worse outcome.
Inflammatory bowel disease questionnaire (IBDQ) | Week 12
  Differences in Inflammatory Bowel Disease Questionnaire (IBDQ) scores from baseline at 12 weeks were used for between-group assessment. The minimum score is 32, and the maximum score is 224. Higher scores mean a better outcome.
Safety evaluation (number of participants with abnormal routine blood tests) | Week 12
  Routine blood tests, which mainly include the number of red blood cells, white blood cells and platelets per litre of blood.
Safety evaluation (number of participants with abnormal Liver function tests) | Week 12
  Liver function tests, mainly including peripheral blood concentrations of alanine aminotransferase (U/L), glutamine aminotransferase (U/L), gamma-glutamyl transpeptidase (U/L), alkaline phosphatase (U/L), total bilirubin (μmol/L), direct bilirubin (μmol/L), indirect bilirubin (μmol/L), total protein (g/L), albumin (g/L) and globulin (g/L).
Safety evaluation (number of participants with abnormal Renal function tests) | Week 12
  Renal function tests, mainly including tests of creatinine (μmol/L) and urea nitrogen (mmol/L) concentrations in peripheral blood.

OTHER OUTCOMES:
Gut microbiota composition structure and function | Week 12
  Differences in the compositional structure and function of the intestinal flora in CD patients with abdominal pain before and after 12 weeks of acupuncture treatment.
Correlation between changes in relative abundance of gut microbes and abdominal pain | Week 12
  Correlation between the relative abundance data of intestinal microbiota which analyzed by metagenomics at different taxonomic levels, such as Phylum,Class,Order,Family, and changes in of abdominal pain VAS score before and after 12 weeks of acupuncture treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, PhD, MD, Study Chair — Shanghai Institute of Acupuncture, Moxibustion and Meridian
Locations (1):
- Shanghai Institute of Acupuncture, Moxibustion and Meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: No